CLINICAL TRIAL: NCT00005795
Title: Phase II Trial of Arsenic Trioxide in Relapsed and Refractory Acute Myeloid Leukemia, Secondary Leukemia, and/or Newly-Diagnosed Patients Greater Than or Equal to 65 Years Old
Brief Title: Arsenic Trioxide in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NCI 99H6; NU-99H6; NU-476-016; NCI-T99-0094
Record Dates: First submitted 2000-06-02; First posted 2004-02-16 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); secondary acute myeloid leukemia; adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the rate of response (complete or partial remission), duration of response, relapse free survival, and overall survival of patients with relapsed or refractory acute myeloid leukemia (AML) or untreated older patients or those with secondary AML when treated with arsenic trioxide. II. Evaluate the toxicities of this agent in this patient population. III. Measure degree of apoptosis induced and/or differentiation in pretreatment and posttreatment AML cells.

OUTLINE: Patients receive arsenic trioxide IV over 1-4 hours daily for up to 60 days, or until bone marrow blasts are less than 5%, followed by 4-6 weeks of rest. After the first course, additional courses of arsenic trioxide last 25 days. Treatment continues for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients with a complete response (CR) receive 1 additional 25 day course after achieving CR. Patients are followed monthly for 6 months, every 2 months for 6 months, every 3 months for 12 months, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 12-35 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Documented acute myelogenous leukemia (AML) including secondary AML and biphenotypic leukemia Secondary AML may be either chemotherapy induced or evolving from a myelodysplastic syndrome Bone marrow evidence of AML must include the following: Cellularity of 20% or greater Minimum of 20% leukemic cells Signs of bone marrow failure such as: Anemia (hemoglobin less than 12.0 g/dL) Granulocytopenia (granulocyte count less than 1,500/mm3) Thrombocytopenia (platelet count less than 100,000/mm3) Must not be any of the following: Acute lymphoblastic leukemia Blastic phase of chronic myelogenous leukemia Acute promyelocytic leukemia (M3) Prior induction therapy using any conventional induction chemotherapy regimen required In first or second relapse after successful induction therapy OR Failed 1 attempt at reinduction relapse OR Refractory to at least 1 prior induction therapy No prior induction therapy allowed in secondary AML or in newly diagnosed AML in patients at least 65 years old

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-2 Life expectancy: At least 6 weeks Hematopoietic: See Disease Characteristics No evidence of being platelet transfusion refractory WBC no greater than 20,000/mm3 (leukapheresis, hydroxyurea, or both allowed) Hepatic: Bilirubin no greater than 2.0 mg/dL unless leukemic infiltration to liver SGOT or SGPT less than 2 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No evidence of symptomatic coronary atherosclerotic heart disease Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception No active infection and afebrile Afebrile, stable, and completing antibiotics allowed Febrile not from infection but from blood products allowed

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent bone marrow transplantation Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: No other concurrent antileukemic agents

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2000-02; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin S. Tallman, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States